CLINICAL TRIAL: NCT04694079
Title: VOYAGE- Ventricular Tachycardia Ablation and Myocardial Scar Characterization With Magnetic Resonance
Brief Title: Ventricular Tachycardia Ablation and Myocardial Scar Characterization With Magnetic Resonance
Acronym: VOYAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Collaborators: Azienda USL Toscana Nord Ovest (Other); Azienda USL Toscana Sud Est (Other Government); Azienda Ospedaliera Universitaria Senese (Other); Fondazione Toscana Gabriele Monasterio (Other); Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Giulio Zucchelli, Principal investigator, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17288
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Ventricular Tachycardia; Myocardial Fibrosis
Keywords: Ventricular tachycardia; Cardiac magnetic resonance; Cardiac ablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, multicentric open-label study with control group. Superiority of VT ablation including myocardial scar characterization (group 1+2) in comparison with only EAM-guided ablation (group 3: control) in terms of 12-months freedom of recurrences, will be evaluated as primary hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1, CMR-guided VT ablation (Experimental): Patients randomized to Group 1, will undergo CMR-guided VT ablation. LGE-CMR data obtained by 1,5 or 3 T CMR and multi-detector cardiac tomography (MDCT) data obtained using a 128 slice CT scanner will be processed with ADAS-VT software (Galgo Medical, Barcelona, Spain).
  Ablation procedure will be carried out in an electrophysiology lab by using the CARTO 3 electroanatomical mapping system (Biosense Webster, Diamond Bar, CA, USA). A ThermoCool SmartTouch SF open irrigated 3,5 mm tip radiofrequency catheter (Biosense Webster, Diamond Bar, CA, USA) will be used both for mapping and ablation.
  Interventions: Procedure: Group 1, CMR-guided/aided VT ablation
- Group 2, CMR-aided VT ablation (Experimental): Patients randomized to Group 2, will undergo CMR-aided VT ablation. LGE-CMR data obtained by 1,5 or 3 T CMR and multi-detector cardiac tomography (MDCT) data obtained using a 128 slice CT scanner will be processed with ADAS-VT software (Galgo Medical, Barcelona, Spain).
  Ablation procedure will be carried out in an electrophysiology lab by using the CARTO 3 electroanatomical mapping system (Biosense Webster, Diamond Bar, CA, USA). A ThermoCool SmartTouch SF open irrigated 3,5 mm tip radiofrequency catheter (Biosense Webster, Diamond Bar, CA, USA) will be used both for mapping and ablation.
  Interventions: Procedure: Group 2, CMR-aided VT ablation
- Group 3, Electroanatomical guided ablation (Active Comparator): Patients assigned to Group 3, will not undergo LGE-CMR. Ablation procedure will be carried out in an electrophysiology lab by using the CARTO 3 electroanatomical mapping system (Biosense Webster, Diamond Bar, CA, USA). A ThermoCool SmartTouch SF open irrigated 3,5 mm tip radiofrequency catheter (Biosense Webster, Diamond Bar, CA, USA) will be used both for mapping and ablation.
  Interventions: Procedure: Group 3, Electroanatomical guided ablation

INTERVENTIONS:
Procedure: Group 1, CMR-guided/aided VT ablation — Ablation of the "anatomical" channels of heterogeneous tissue within the scar
  Arms: Group 1, CMR-guided VT ablation
Procedure: Group 2, CMR-aided VT ablation — Ablation of the "electrical" conduction channels within the scar
  Arms: Group 2, CMR-aided VT ablation
Procedure: Group 3, Electroanatomical guided ablation — Ablation guided by an electro-anatomical system without the aid of CMR
  Arms: Group 3, Electroanatomical guided ablation

SUMMARY:
Previous monocentric experiences have already highlighted the role of preoperative cardiac imaging, in particular of cardiac magnetic resonance (CMR) and tomography (CT), in improving the ablation results of scar-related ventricular tachycardia (VT). A better characterization of scar obtained with high quality CMR images and post processing data with creation of maps exploring the heart in concentric layers from the endocardium to the epicardium could allow a personalized and more precise approach to this pathology.

Aim of the study - Evaluating the feasibility and possible benefit of CMR-guided ablative approach (group 1: ablation of the "anatomical" channels of heterogeneous tissue within the scar) compared to CMR-aided approach (group 2: ablation of the "electrical" conduction channels within the scar) and standard approach (group 3: ablation guided by an electro-anatomical system without the aid of CMR) in a multi-center Tuscan study.

What would add the project to what is known - The achievement of the objectives by the project would allow to propose a personalized ablation on the basis of the scar characterization and would allow a better efficacy, efficiency of the procedure and probably also a safer treatment

DETAILED DESCRIPTION:
State of the art and preliminary data

Patients with structural heart disease (SHD) are at increased risk of VAs that can promote life-threatening events, for whom a proper treatment has a pivotal role. The use of antiarrhythmic drugs is limited due to their ineffectiveness in reducing related mortality or their common side effects. Implantable cardioverter defibrillator (ICD) can improve survival in a certain group of patients with SHD, but recurrent ventricular tachycardia (VT) needing ICD shocks reduce quality of life and probably patients survival. Moreover, ICD implant is affected by a noticeable risk of acute and chronic complications, that can reduce the survival of ICD recipient. Catheter ablation is an effective technique especially for the management of post-myocardial infarction ventricular tachycardia (post-myocardial infarction VT) and the recent VANISH trial showed that ablation reduced the composite primary outcome of death, VT storm or appropriate ICD shocks compared to patients with an escalation of amiodarone.

The introduction of a catheter in the ventricular chambers through a vascular access, allows to map the VT circuit that is usually inside the scar, and perform an ablation of the tissue responsible of the VAs substrate. The signals recorded by the catheter and the fluoroscopy images have been used to localize the target since 90s, but in the last decade the emergence of technological innovations, such as three-dimensional electroanatomic mapping (3D-EAM), has enhanced our ability to identify ablation targets. Three-dimensional electroanatomic mapping enables to generate a 3D reconstruction of any part of the heart without needing fluoroscopic navigation. Integration between anatomic and electrocardiographic (ECG) data it is very useful in choosing an optimal location for VA ablation, and the use of mapping systems contributed to reduce procedural, fluoroscopy and radiofrequency time. However, the efficacy of 3D-EAM can be suboptimal when we decide to follow a strategy of substrate ablation. Substrate ablation is characterized by an ablation of abnormal electrograms (EGMs) identified during sinus rhythm or ventricular pacing. In a recent meta-analysis, the combined risk of ventricular arrhythmia recurrence and all-cause mortality during long-term follow-up was lower when using a substrate-based approach compared to standard ablation of stable VT. However, efficacy was greatly reduced if the homogenization of the arrhythmic substrate was incomplete.

Real-time integration of anatomical VT substrate from data coming from cardiac image such as cardiac magnetic resonance (CMR) and multidetector computed tomography (CT) with EAM seems to improve efficacy of VA radiofrequency ablations and use of scar integration from imaging was an independent predictors of VT-free survival after catheter ablation in post-MI VT in recent papers. However, integration of CMR and CT images in the EAM system hasn't allowed to avoid, until now, an EAM that is time consuming, often imprecise and allowing only an incomplete substrate modification. Based on this consideration, we thought that an image integration taking into account not only the location of scar, but also its quantification and characterization could increase the efficiency of the ablation procedure, with an improvement of acute and chronic outcome. For this purpose, CMR has a pivotal role, allowing at characterizing the scar tissue via color-coded pixel signal intensity (PSI) maps that have a high correlation with the electroanatomic maps obtained during the ablation procedures. Particularly, the VT isthmuses found with the EAM correlated with the presence of heterogeneous tissue channels (HTCs) depicted in the PSI maps. Previous experiences demonstrated that these PSI maps can be imported in the navigation system to help substrate ablation, but only if they are obtained from high spatial resolution late gadolinium enhancement (LGE)-CMR images. One recent publication showed that CMR-aided scar dechanneling was associated with a lower need for ablation delivery, higher non-inducibility rates after substrate ablation, and reduced VT recurrences in the follow-up. In brief, in this experience the target ablation sites were the conducting channels (CC) entrances (i.e. entrances of VT isthmuses) identified in the substrate EAM, but PSI maps integrated into the navigation system were used to focus on specific regions of the scar. The authors found 23% of false negative (CCs evidence outside the HTCs entrances) and 16% of false positives (HTCs only identified in PSI maps). The HTCs identified only in the PSI maps, without matching with a CC on the EAM, were not targeted for ablation. Very recently, the same group presented results about a possible improvement of the outcome (particularly the efficiency, but probably with extension to efficacy and safety) using a CMR guided ablation, targeting only the HCTs (all of them). However, both experiences with CMR aided and guided ablation had been performed with a retrospective design and in a single-centre high volume laboratory, and for this reason we don't know the potential application of this technique in the real world of clinical electrophysiology.

The investigators sought to evaluate the feasibility, efficacy, safety and efficiency of a VT ablation guided or aided by CMR in comparison with VT ablation guided only by EAM (standard approach nowadays).

General goal of the Project

The project aims at developing a network between Tuscany centres for scar-related VT ablation, based on an accurate patients' selection, an anatomic substrate definition with radiomics, a qualitative analysis of the radiomic data via an artificial intelligence with a cardiac shell reconstruction that will be used in the electrophysiological laboratory to tailor a specific and personalized ablation procedure. To test whether this tailored approach could improve our clinical approach we built the following experimental design. Briefly, patients with VT arriving at each hospital of the consortium from either emergency room, outpatient clinic, or other hospitals, will be evaluated for SHD. Patients with confirmed diagnosis of SHD can be enrolled in the study and will be further evaluated to determine whether there are no contraindications to CMR. If they have contraindications to CMR or CMR images are suboptimal the patients will undergo EAM-guided VT ablation, vice versa they will be randomized to a CMR-guided or -aided ablation. Data obtained from LGE-CMR will be processed with the ADAS-VT software (Galgo Medical, Barcelona, Spain), an artificial intelligence suite used to create a 3D multi-layer map of the ventricular wall.

At the end, the patients will be divided in 3 groups:

* Group 1: patients undergoing CMR guided VT ablation (ablation focused only on HTCs)
* Group 2: patients undergoing CMR aided VT ablation (ablation focused only on CCs on EAM, but with integration of CMR derived shell in the map and with scar projection (with HTCs on the EAM)
* Group 3 (control): patients with contraindication to CMR (or poor-quality images deemed unsuitable for further analysis) undergoing EAM-guided VT ablation without any CMR data about scar (core and border zone)

Aim of the study

Evaluating the feasibility and possible benefit of CMR-guided ablative approach (group 1: ablation of the "anatomical" channels of heterogeneous tissue within the scar) compared to CMR-aided approach (group 2: ablation of the "electrical" conduction channels within the scar) and standard approach (group 3: ablation guided by an electro-anatomical system without the aid of CMR) in a multi-centre Tuscan study.

Primary objective (see after)

Secondary objective (see after)

Study design (see after)

Population of the study

103 patients with VT in patients with SHD will be recruited in 7 Tuscan hospitals participating in the project.

Study setting

Regional network of hospitals including tertiary centres with an electrophysiology team of qualified investigators/physicians with proven experience in performing ventricular tachycardia ablation.

Inclusion Criteria (see after)

Exclusion Criteria (see after)

Withdrawal from the study

* Informed consent withdrawal
* Patients enrolled without satisfied inclusion criteria or in presence of exclusion criteria

Acute Procedure endpoints Acute success will be defined as non-inducibility of any sustained monomorphic VT at the end of the procedure. Partial success will be considered with the clinical VT successfully ablated with other monomorphic VTs remaining inducible. Pre-ablation inducibility is not be required.

Device programming

All patients involved in the study, regardless of Group allocation, will have their ICD programmed following 2019 HRS/EHRA/APHRS/LAHRS expert consensus statement on optimal ICD programming, following the manufacturer specific recommendations about therapy and detection in patients where VT cycle is known, alongside any anti-bradycardia setting necessary for therapeutic needs. Particularly, the VT zone with lower rate detection should be set at 10-20 ipm slower than the clinical VT to guarantee a good sensitivity in recurrences diagnosis and therapy should be programmed in order to reduce unnecessary shocks. 26

Medical therapy

Patients involved in the study will be treated with antiarrhythmic drugs and any other medical therapy considered standard of care for the SHD and VT. Particularly, use of amiodarone is allowed at enrollment but is strongly suggested to stop it at 1 month follow-up, if not contraindicated, to avoid drug-related toxicity and not to confound trial results about primary objective.

Potential risks

No extra risks appear to be related to study participation. Risks are related to the procedure itself, which is explained on the informed consent sheet.

Potential benefits

Thanks to preprocedural CMR imaging, patients assigned to both interventional groups (1 and 2) could benefit from potentially shorter procedures and lower radiological exposure with shorter fluoroscopy time. Patients assigned to Group 2 will benefit from an overall shorter EAM acquisition phase, given the fact that the area of interest will be determined by CMR-LGE data. Due to the complete absence of EAM, patients assigned to Group 1 could benefit from even smaller procedural time and radiological exposure.

Moreover, patients assigned to CMR-guided ablation (group 1) and CMR-aided ablation (group 2) could benefit from improved VT substrate identification. CMR-derived PSI maps could improve CC entrance localization compared to the standard technique based on the voltage map obtained from EAM. We anticipate that improved scar definition and CC entrance localization could lead to a significant improvement in substrate elimination, and, ultimately, to better acute and long-term outcomes. The ablation at HTCs entrance in group 1 could improve acute efficacy compared to the other groups, as showed by recent unpublished data (Soto Iglesias et al. JACC EP 2020).

Study conclusion

The study will conclude with the 12-months follow-up of the last enrolled patients (see sample size), and each patient with 12-months follow-up will exit from the study. Patients will have the possibility to exit from the study at any time they decide without any explanation about it. Principal investigator will have the ultimate authority to stop the trial at any time of enrollment if any harms emerge during trial conduction. Once the study is completed, principal investigator or delegate will notify the site of closeout and a study closeout visit will be performed.

Study endpoint (see after)

Procedural evaluation

Any variables evaluated as study endpoint (see above) will be collected.

Quality of life assessment

To evaluate potential differences between different interventional approaches in health-related quality of life changes, the 36-Item Short Form Survey (SF-36) will be administered at baseline (before ablation) and at the 12-months follow up visit.

Follow-up

Clinical follow-up (FU) will include outpatient clinic visits at 1, 6 and 12 months after the ablation procedure. If no contraindications, amiodarone (if used) should be stopped at the 1-month FU visit.

At all follow up visits, the following parameters and information will be taken:

* Physical examination
* 12 lead surface ECG
* Transthoracic echocardiography (at 6 and 12 months)
* ICD interrogation, analyzing any event marked as VT or VF by the device.

VT recurrence will be defined as any documented sustained VT (more than 30 s) or appropriate ICD therapy at ICD check.

To assess changes in health-related quality of life, the 36-Item Short Form Survey (SF-36) will be administered at the 12-months follow up visit.

Sample size To test the primary hypothesis, 103 patients will be necessary with 80% power and 5% type 1 error, considering 50% of group 1-2 (low risk), 50% of group 3 (high risk), 16% of likelihood of VT recurrences at 12 months in low risk patients and 44% of likelihood in high risk patients with HR (high risk/low risk of recurrences ) of 2,75 (Cox PH, 2 sided equality).

Screening phase

All patients referred to or directly evaluated at one of the participating centres for VT will be screened for ablation and for study participation. The presence of structural heart disease will be evaluated on the basis of past medical history and available imaging carried out during patient evaluation, such as echocardiography, cardiac CT, or previous CMR.

Enrollment procedure - Recruitment and agenda

All participant centres are referral centres for VT ablation within their health care network. All patients who give informed consent for participation and fulfill the inclusion eligibility criteria will be consecutively enrolled. We expect to include all the patients within a 2-years period. The 12-month follow-up information of the last included patient should be available approximately 3 years after the first inclusion. A monthly assessment of screening database will be performed in order to increase the enrollment procedure.

Group allocation

Patients deemed suitable for CMR according to comorbidities, device MRI-compatibility and willingness to undergo the examination, will be randomly allocated to groups 1 and 2. Patients eligible to join the study but unsuitable for CMR or with poor CMR images will be assigned to Group 3.

Randomization

Randomization will be performed in patients undergoing CMR (Groups 1 and 2) in 1:1 fashion using the app "Randomizer for Clinical Trial Lite" or equivalent web-based platform. The scientific coordinator of the study or a delegate should be the unique responsible of randomization and will be contacted upon all new recruitments.

Blindness

Blindness of patients is not required.

Study procedures

Routine baseline analysis, clinical visit, 12 lead ECG, transthoracic echocardiography, transoesophageal echocardiography, cardiac CT, CMR (if possible), VT ablation. Patients will be hospitalized for the ablation procedure and may undergo any clinical, imaging or lab examination considered necessary for clinical management during their stay.

Data collection

The principal investigator or delegate is responsible of the data collection on the electronic Case Report Forms (eCRFs). The principal investigator or delegate will review all the data on the eCRFs and will sign to verify he has reviewed the data collected. Original anonymized paper support forms will be stored in a secure place and manner at each participating centre. Anonymization codes will be stored in a safely manner by the local principal investigator. Access to the online study data (eCRFs) will be restricted through passwords. In addition, centre coordinators will only have access to their own centre's data. Paper files will be physically stored until 5 years after the completion of the study

Data management

Source documents shall be created and maintained by the investigation site team throughout the clinical investigation. The data reported on the eCRFs shall be derived from, and be consistent with, these source documents, and any discrepancies shall be explained in writing. The eCRFs shall be signed and dated by the principal investigator or a delegated investigator. Any change or correction to data reported on a paper CRF shall be dated, initialed and explained if necessary, and shall not obscure the original entry.

Traceability of documents and data

The investigator shall ensure accuracy, completeness, legibility and timeliness of the data reported to the principal investigator on the eCRFs and in all required reports. When copies of the original source document as well as print outs of original electronic source documents are retained, these shall be signed and dated by a member of the investigational site team with a statement that it is a true reproduction of the original source document.

Protocol deviation

A protocol deviation is defined as a situation in which there is a non-compliance with the protocol. The following situations are considered protocol deviations and must be appropriately documented:

1. Patient assigned to Group 1 or 2 and with a good quality CMR is not treated in his predefined group.
2. Patient assigned to control group undergo good quality CMR, which is used to plan ablation strategy.
3. Patient assigned to control group undergo good quality CMR and eventually a CMR-guided or aided ablation.
4. Amiodarone is not discontinued at 1 month Follow-up.
5. ICD is not programmed following guidelines, as previously stated.
6. Patient without SHD, or in presence of other exclusion criteria, is enrolled in the study.

Investigators will be required to adhere to the investigational plan, signed investigator's agreement, applicable national or local, laws and regulations, and any conditions required by the appropriate Ethics Committees or applicable regulatory authorities. The reporting of all the deviations will be performed through the electronic case report form (e-CRF) application. In the event of repeated protocol deviation as determined by the principal investigator, a clinical research associate or clinical representative will attempt to secure compliance by one or more of the following actions: 1) contacting the investigator by telephone, or 2) contacting the investigator in writing.

Statistics

All applicable statistical tests will be 2-sided and will be performed using a 5% significance level. Continuous variables will be reported as mean ± standard deviation, or median (range or interquartile range if data are skewed) if not normally distributed; these variables will be compared using Student's t-test if normally distributed, Aspin-Welch test if normally distributed with unequal variance demonstrated using Variance-ratio F-test, or Mann-Whitney U test if not normally distributed. Categorical variables will be expressed as total number (percentage) and will be compared by chi-squared test. As far as the primary endpoint, data will be analyzed according to the intention-to-treat principle. Survival free from ventricular arrhythmia, will be evaluated using a time-to-first-event analysis with the Logrank test and the Kaplan-Meier cumulative event rate. A multivariable Cox proportional hazards model will be performed to investigate the effects of baseline characteristics in predicting ablation results.

Event definitions

Adverse event: any untoward medical occurrence in a clinical trial participant that does not necessarily have a causal relationship with the treatment.

Adverse reaction: any untoward or unintended response to an investigational therapy.

Serious adverse event: any untoward medical occurrence that

* Results in death
* Is life-threatening
* Requires inpatient hospitalization or causes prolongation of existing hospitalization
* Results in persistent or significant disability/incapacity,
* May have caused a congenital anomaly/birth defect, or
* Requires intervention to prevent permanent impairment or damage.

Event registration and causal relationship

All adverse events judged by an investigator as having a reasonal possibility of a causal relationship to an investigational therapy would qualify as an adverse reaction. The expression "reasonable causal relationship" means to convey, in general, that there is evidence or argument to suggest a causal relationship.

Event reporting

Any adverse event will be stored in the eCRF and reported to the principal investigator, the local Institution Review Board and the Ethics Committee according to the ICH Guideline for Clinical Safety Data Management and the 2016 EMA/CHMP/ICH/135/1995 Guideline for good clinical practice E6(R2).

Funding

The project will receive government funding from the only sponsor Regione Toscana according to the "Bando Ricerca Salute 2018 - D.D n.975, 16/1/2020".

Role of the sponsor (Tuscan region)

According to Regional Law 20/2009 the research project has already undergone initial evaluation and approval by the sponsor and will undergo further scrutiny during the preliminary phase, during enrollment and after study completion. Technical financial reports will be filed to the sponsor mid-enrollment and upon study completion.

The sponsor will not play any role in patient selection and trial management.

Insurance

A Trials insurance will provide protection for the sponsors/organisers of clinical trials, covering their legal liability to pay compensation in the event of an injury to a trial participant. The coverage of insurance cost is included in the budget of the funding received from the sponsor.

Review of data

The clinical investigation will be monitored by reviewing the e-CRF submitted by the investigators. The following activities will occur:

* All e-CRFs will be reviewed for completeness and accuracy upon receipt by the principal investigator or delegate.
* The investigator (co-investigator) and/or delegate will be contacted by the principal investigator regarding any missing or unclear data.

An interim analysis will be conducted after 12 month since the first patient enrollment to evaluate the enrollment rate, the initial results and other factors which reflect the overall progress and integrity of the study.

Clinical committee for Data Monitoring

The monitoring of data accuracy will be performed by principal investigator or delegate as previously stated (see review of data). No external clinical committee are considered for this task.

Protocol amendments

Any modifications to the protocol which may impact on the conduct of the study, potential benefit of the patient or may affect patient safety, including changes of study objectives, study design, patient population, sample sizes, study procedures, or significant administrative aspects will require a formal amendment to the protocol. Any amendment to the protocol will be notified to the Ethical Committee, to the sponsor and to all participating centres.

Ethics and Disseminations

This protocol is in line with the standard ethic principles for clinic research and good clinical practice according to the ICH Guideline for Clinical Safety Data Management and the 2016 EMA/CHMP/ICH/135/1995 Guideline for good clinical practice E6(R2), and must be reviewed and approved by the local institutional review board (IRB) of each centre.

Informed consent form

Any subject admitted as outpatient or inpatient at one the participating centres diagnosed with VT will be scrutinized for study participation. Patients deemed suitable to join the trial according to eligibility criteria will be asked informed consent for study enrolment. Patients willing to participate and diagnosed with SHD will be assigned to a Group according to protocol. Patients under 18 will not be screened according to eligibility criteria. Patients permanently or temporarily lacking legal capacity will not be screened. Patients eligible to join an interventional Group (1 and 2) will be randomized within 1 month since study enrolment.

Confidentiality

All study-related information will be stored securely at the study site up to 7 years after the end of the study. All participant information will be stored in locked file cabinets in areas with limited access. All laboratory specimens, reports, data collection, process, and administrative forms will be identified by a coded ID number only to maintain participant confidentiality. All records that contain names or other personal identifiers, such as locator forms and informed consent forms, will be stored separately from study records identified by code number. All local databases will be secured with password-protected access systems.

Conflicts of interest

Dr. Berruezo is a stockholder in Galgo Medical SL and has received financial support from Siemens Healthcare. The other authors have no other relevant affiliations or financial involvement with any organization or entity with a financial interest in or financial conflict with the subject matter or materials discussed in the study apart from those disclosed.

After beginning of the project and financial coverage by the Tuscany region, other investigators will be defined (personnel with fixed-term employment relationships specifically hired for the project) for data management, study monitoring and Core Lab institution.

Data property

Project Principal Investigators will have direct access to their own site's data sets and may access to other sites' data only by request. To ensure confidentiality, data dispersed to project team members will be blinded of any identifying participant information.

Dissemination policy

The study results will be released to the participating physicians, referring physicians, patients and the general medical community during medical congresses or through publication, expected after the end of follow-up. The principal investigator of the coordinating centre of the study will take the decision to submit the report for publication and will have ultimate authority over all the activities.

ELIGIBILITY:
Inclusion Criteria:

* Indication for VT ablation in patients with SHD (indications according to the 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death);
* Structural heart disease (clinical history, EKG, multimodality imaging)
* Signed informed consent;

Exclusion Criteria:

* Age <18 y;
* ICD not already implanted nor expected within 1 month;
* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons);
* Inability to give written informed consent;
* Pregnancy (suspected or confirmed);
* Acute coronary syndrome in the previous 3 months;
* Creatinine clearance < 15 ml/min (stage 5 CKD) (according to clinical history or out/in-patient tests performed upon enrollment)
* Severe chronic liver disease (Child-Pugh score C) (according to clinical history or out/in-patient tests performed upon enrollment)
* Heart surgery for valve disease in the previous 6 months or expected within 6 months,
* NYHA functional class IV heart failure or CCS functional class IV angina
* Previous VT ablation (redo procedure).
* Systemic illness likely to limit survival to < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
VT recurrences | 12-month
  To compare the recurrences of the CMR guided/aided approaches in comparison to control group

SECONDARY OUTCOMES:
Efficiency | 1 month
  To evaluate the efficiency (procedure times, radiofrequency time, fluoroscopy time) of different approaches
VT non-inducibility | 1 month
  To evaluate the VT non-inducibility of different approaches at the end of ablation
Number of participants with Complications | 12-month
  To compare the Number of participants with Complications using a CMR-guided/aided approach in comparison with control group
Rate of ICD interventions | 12-month
  To compare the outcome of the CMR guided/aided approaches of VT ablation in terms of ICD interventions rate per patients with recurrences (ATP or shocks) during 12 months follow-up in comparison to control group
CMR images suitability | 1 month
  To evaluate the possibility to use the CMR images for a CMR-guided/aided approach (rate of patients who had underwent CMR, in whom the images are suitable for a CMR guided/aided approach)

CONTACTS AND LOCATIONS:
Overall Officials: GIULIO ZUCCHELLI, MD, PhD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (7):
- Italy (7):
  - Azienda USL Toscana Sud Est, Arezzo, AR
  - Azienda USL Toscana Sud Est- U.O.C. Cardiologia, Ospedale Misericordia - Grosseto, Grosseto, GR
  - Azienda USL Toscana Nord Ovest- U.O.C. Cardiologia, Ospedali Riuniti - Livorno, Livorno, LI
  - Azienda USL Toscana Nord Ovest - U.O.C. Cardiologia, Ospedale Versilia, Camaiore, LU
  - AOUPisana, Pisa, PI
  - FTGM, Pisa, PI
  - Azienda Ospedaliero Universitaria Senese - U.O.C. Cardiologia, Siena, Siena, SI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Blom N, Borggrefe M, Camm J, Elliott PM, Fitzsimons D, Hatala R, Hindricks G, Kirchhof P, Kjeldsen K, Kuck KH, Hernandez-Madrid A, Nikolaou N, Norekval TM, Spaulding C, Van Veldhuisen DJ; ESC Scientific Document Group. 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: The Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC). Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC). Eur Heart J. 2015 Nov 1;36(41):2793-2867. doi: 10.1093/eurheartj/ehv316. Epub 2015 Aug 29. No abstract available. PMID 26320108
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Soto-Iglesias D, Acosta J, Penela D, Fernandez-Armenta J, Cabrera M, Martinez M, Vassanelli F, Alcaine A, Linhart M, Jauregui B, Efimova E, Perea RJ, Prat-Gonzalez S, Ortiz-Perez JT, Bosch X, Mont L, Camara O, Berruezo A. Image-based criteria to identify the presence of epicardial arrhythmogenic substrate in patients with transmural myocardial infarction. Heart Rhythm. 2018 Jun;15(6):814-821. doi: 10.1016/j.hrthm.2018.02.007. Epub 2018 Feb 7. PMID 29427821
- [Background] Andreu D, Ortiz-Perez JT, Fernandez-Armenta J, Guiu E, Acosta J, Prat-Gonzalez S, De Caralt TM, Perea RJ, Garrido C, Mont L, Brugada J, Berruezo A. 3D delayed-enhanced magnetic resonance sequences improve conducting channel delineation prior to ventricular tachycardia ablation. Europace. 2015 Jun;17(6):938-45. doi: 10.1093/europace/euu310. Epub 2015 Jan 23. PMID 25616406
- [Background] Soto-Iglesias D, Butakoff C, Andreu D, Fernandez-Armenta J, Berruezo A, Camara O. Integration of electro-anatomical and imaging data of the left ventricle: An evaluation framework. Med Image Anal. 2016 Aug;32:131-44. doi: 10.1016/j.media.2016.03.010. Epub 2016 Apr 4. PMID 27086166
- [Background] Porras AR, Piella G, Berruezo A, Fernandez-Armenta J, Frangi AF. Pre to Intraoperative Data Fusion Framework for Multimodal Characterization of Myocardial Scar Tissue. IEEE J Transl Eng Health Med. 2014 Sep 4;2:1900211. doi: 10.1109/JTEHM.2014.2354332. eCollection 2014. PMID 27170873
- [Background] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033
- [Background] Yamashita S, Cochet H, Sacher F, Mahida S, Berte B, Hooks D, Sellal JM, Al Jefairi N, Frontera A, Komatsu Y, Lim HS, Amraoui S, Denis A, Derval N, Sermesant M, Laurent F, Hocini M, Haissaguerre M, Montaudon M, Jais P. Impact of New Technologies and Approaches for Post-Myocardial Infarction Ventricular Tachycardia Ablation During Long-Term Follow-Up. Circ Arrhythm Electrophysiol. 2016 Jul;9(7):e003901. doi: 10.1161/CIRCEP.116.003901. PMID 27406604
- [Background] Piers SR, Tao Q, de Riva Silva M, Siebelink HM, Schalij MJ, van der Geest RJ, Zeppenfeld K. CMR-based identification of critical isthmus sites of ischemic and nonischemic ventricular tachycardia. JACC Cardiovasc Imaging. 2014 Aug;7(8):774-84. doi: 10.1016/j.jcmg.2014.03.013. Epub 2014 Jul 16. PMID 25051947
- [Derived] Lilli A, Parollo M, Mazzocchetti L, De Sensi F, Rossi A, Notarstefano P, Santoro A, Aquaro GD, Cresti A, Lapira F, Faggioni L, Tessa C, Pauselli L, Bongiorni MG, Berruezo A, Zucchelli G. Ventricular tachycardia ablation guided or aided by scar characterization with cardiac magnetic resonance: rationale and design of VOYAGE study. BMC Cardiovasc Disord. 2022 Apr 14;22(1):169. doi: 10.1186/s12872-022-02581-1. PMID 35421939